CLINICAL TRIAL: NCT02754843
Title: Quality Control of CE-Labelled Phonak Hearing Systems (Study Part: Sonova2015-00)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: Sonova2015-00
Record Dates: First submitted 2015-10-16; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Naida Q90-SP (Active Comparator): Phonak's commercial power Behind-The-Ear (BTE) device, type 1.
  Interventions: Device: Phonak's equivalent newly developped power BTE; Device: Equivalent competitor device
- Naida Q90-UP (Active Comparator): Phonak's commercial power Behind-The-Ear (BTE) device, type 2.
  Interventions: Device: Phonak's equivalent newly developped power BTE; Device: Equivalent competitor device

INTERVENTIONS:
Device: Phonak's equivalent newly developped power BTE
Device: Equivalent competitor device

SUMMARY:
The purpose of this study, which contains a series of successive study parts, is to methodically evaluate Phonak Hearing Systems on hard of hearing participants to grant quality control prior to each product launch.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impaired persons with and without (experience with) hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the medical device in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility in quiet. Discrimination [%] | One week.
  The data, serving as primary outcome, are collected in a series of lab appointments. The speech intelligibility in quiet will be assessed with the aid of the German rhyme test "Einsilber-Reimtest nach von Wallenberg und Kollmeier" (WaKo). The result is the speech intelligibility in percent. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Speech intelligibility in noise. Speech Reception Threshold [dB SNR] | One week.
  The data, serving as primary outcome, are collected in a series of lab appointments. The speech intelligibility in noise will be assessed with the aid of the German Oldenburger sentence test. The result is the Speech Reception Threshold [dB SNR]. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

SECONDARY OUTCOMES:
Phoneme Perception Test, test no. 1. | Four weeks
  Free field audiometry using narrow band high frequency signals to measure detection thresholds [dB]. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Phoneme Perception Test, test no. 2. | Four weeks
  Free field audiometry using high frequency phonemes to capture their recognition thresholds [dB]. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Phoneme Perception Test, test no. 3. | Four weeks
  Free field audiometry using high frequency phonemes to capture the subjects' distinction capabilities [confusion matrix]. Descriptive statistics will be executed in the form of determining the median and quartiles. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Diary to describe hearing impressions in everyday life | Six weeks
  Subjects are asked to describe their subjective experiences in different listening situations, in daily life, with the aid of quantitative questionnaires. the results are "Yes/No" replies and open-ended.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ebbing, B.Sc., Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Canton Zürich, Switzerland